CLINICAL TRIAL: NCT04829474
Title: Descriptive Factors of Intimate Partner Violence on Women Related to "Incapacité Totale de Travail" : Multicenter Prospective Study
Brief Title: Severe Women Injury Factors Test (SWIFT)
Acronym: SWIFT
Status: Terminated | Type: Observational
Why Stopped: recruitment is insufficient and the current context does not allow satisfactory data collection
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Other Study IDs: CHRO-2021-02
Record Dates: First submitted 2021-03-31; First posted 2021-04-02 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Spouse Abuse
Keywords: Intimate partner violence; Descriptive factors; "Incapacité Totale de travail"
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women consulting for spouse abuse: The study focuses on women consulting a doctor as part of spouse abuse, whatever the context (at the request of the police or not) or their motivation (medical or social).
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — It is a survey that the patient and doctor must complete.

SUMMARY:
Intimate partner violence is a real public health problem, and affects all socio-cultural backgrounds It is defined by behavior within an intimate relationship that causes physical, psychological or sexual harm or suffering to the people in that relationship.

Several risk factors exist such as young age, low level of education, exposing to violence during childhood, pregnancy or addictions.

DETAILED DESCRIPTION:
Routine screening is recommended with redaction of medical certificate in which doctor have to determine l'"Incapacité Totale de Travail" corresponding to the duration of discomfort (physical and psychological repercussions) in the activities of daily life.

It is a legal notion allows to rule on the responsibility of the author. The sentence is increased if the ITT is greater than 8 days.

Worldwide, 30% of women suffered violence whose most common form is intimate partner violence, but legal proceedings have been initiated in less than 25% of the cases.

The trauma of women victims of domestic violence worsens with the repetitions of assaults.

The investigators suppose that the duration of ITT is an indicator of the severity of the injuries sustained.

So, the investigators want to highlight the socio-demographic characteristics and describe the spouse abuse, and then related theese factors to " Incapacité Totale de Travail " (term used in law. It is a scale for assessing the importance of injuries).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Admission to emergency for intimate partner violence
* Or consultation to SOS doctor for intimate partner violence
* Or consultation to medico-judicial unit for intimate partner violence
* No verbal opposition to inclusion

Exclusion Criteria:

* Non intimate partner violence
* Patient under guardianship or curatorship
* Non French speaker
* Coma or inability to express non-opposition
* Prior participation in another center

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult women consulting a doctor for intimate partner violence
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-07-23 (Actual); Study Completion 2021-07-23 (Actual)

PRIMARY OUTCOMES:
Descriptive factors of intimate partner violence on women related to "Incapacité Totale de Travail" | Month 24
  Highlight the socio-demographic characteristics and the violence suffered by women victims of intimate partner violence, and related this factors to " Incapacité Totale de travail "

SECONDARY OUTCOMES:
Descriptive factors of intimate partner violence on women related to "Incapacité Totale de travail" for more than eight days. | Month 24
  Highlight the socio-demographic characteristics and the violence suffered by women victims of intimate partner violence, and related this factors to an " Incapacité Totale de travail " for more than eight days.
Spontaneus request of a medical certificate during the consultation. | Month 24
  Determine the proportion of women asking for a medical certificate during the consultation.

CONTACTS AND LOCATIONS:
Overall Officials: Julien PASSERIEUX, Dr, Principal Investigator — CHR d'Orléans
Locations (5):
- France (5):
  - Regional Hospital center of Orleans, Orléans
  - Centre Hospitalier Régional d'Orléans (UMJ), Orléans
  - CHRU de Tours (SAU), Tours
  - CHRU de Tours (UMJ), Tours
  - SOS Médecins Tours, Tours

REFERENCES:
- [Background] Leppakoski T, Paavilainen E, Astedt-Kurki P. Experiences of emergency care by the women exposed to acute physical intimate partner violence from the Finnish perspective. Int Emerg Nurs. 2011 Jan;19(1):27-36. doi: 10.1016/j.ienj.2010.02.006. Epub 2010 May 20. PMID 21193165
- [Background] Saberi E, Eather N, Pascoe S, McFadzean ML, Doran F, Hutchinson M. Ready, willing and able? A survey of clinicians' perceptions about domestic violence screening in a regional hospital emergency department. Australas Emerg Nurs J. 2017 May;20(2):82-86. doi: 10.1016/j.aenj.2017.02.001. Epub 2017 Mar 6. PMID 28279677
- [Background] Lopez-Ossorio JJ, Gonzalez Alvarez JL, Buquerin Pascual S, Garcia LF, Buela-Casal G. Risk factors related to intimate partner violence police recidivism in Spain. Int J Clin Health Psychol. 2017 May-Aug;17(2):107-119. doi: 10.1016/j.ijchp.2016.12.001. Epub 2017 Jan 31. PMID 30487886
- [Background] Lyons VH, Kernic MA, Rowhani-Rahbar A, Holt VL, Carone M. Use of multiple failure models in injury epidemiology: a case study of arrest and intimate partner violence recidivism in Seattle, WA. Inj Epidemiol. 2019 Aug 12;6:36. doi: 10.1186/s40621-019-0215-x. eCollection 2019. PMID 31417842
- [Background] Choi AW, Lo BC, Wong JY, Lo RT, Chau PC, Wong JK, Lau CL, Kam CW. Clinical Features of Heterosexual Intimate Partner Violence Victims With Escalating Injury Severity. J Interpers Violence. 2021 Sep;36(17-18):8585-8605. doi: 10.1177/0886260519850539. Epub 2019 May 29. PMID 31140351